CLINICAL TRIAL: NCT07358481
Title: DEL-DIP: DELphi Procedure for Developing Recommendations for the Implementation of Wearable Devices and Polygenic Risk Scores
Brief Title: DELphi Procedure for Developing Recommendations for the Implementation of Wearable Devices and Polygenic Risk Scores
Acronym: DEL-DIP
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 8217
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Wearable Electronic Devices; Polygenic Risk Score; CVD - Cardiovascular Disease; Primary Prevention
Keywords: cardiovascular prevention
MeSH Terms: conditions — Genetic Risk Score; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- INNOPREV expert panel: Professionals involved in the INNOPREV project with expertise in cardiology, personalized medicine, and/or digital health will be invited to participate. Enrollment will occur by invitation only, contingent upon provision of electronic informed consent. A panel of at least 10 experts is planned

SUMMARY:
DEL-DIP is a prospective observational study employing a Delphi methodology (at least two online rounds) to elicit and consolidate the views of an expert panel within the INNOPREV project. The study aims to develop operational recommendations to support the coordinated implementation of Polygenic Risk Scores (PRS) and wearable devices in cardiovascular prevention. Specifically, it addresses the following research question: which recommendations and requirements-genomic, digital, and clinical/organizational-are necessary to integrate PRS and wearable technologies into routine practice and healthcare services, and for which of these elements do experts achieve consensus (defined as a Content Validity Index, CVI, > 79%)

DETAILED DESCRIPTION:
The DEL-DIP project aims to develop operational recommendations to support the coordinated implementation of Polygenic Risk Scores (PRS) and wearable devices within cardiovascular prevention pathways, where the integration of genomics and digital health may enhance risk stratification and enable continuous monitoring.

The study adopts a Delphi methodology comprising anonymous, web-based rounds in which an expert panel rates its level of agreement with a series of proposed recommendations. Following each round, responses are aggregated and summarized, and the items are re-circulated to allow participants to reconsider and refine their judgments in light of group feedback, thereby facilitating iterative convergence toward consensus.

Data are collected via Microsoft Forms and centralized for analysis. Safeguards are implemented to ensure data security, anonymity, and privacy, and electronic informed consent is obtained prior to questionnaire access.

For each item, the Content Validity Index (CVI) is calculated as the proportion of experts assigning a rating of 4 or 5. A CVI > 79% indicates consensus and supports item inclusion; CVI values between 70% and 79% indicate partial agreement and the need for item revision and/or additional Delphi rounds; values < 70% suggest item exclusion.

The final output will consist of a set of recommendations organized by domain (genomic, digital, and clinical/organizational), together with an assessment of response stability across successive rounds (i.e., changes in CVI), to inform implementation within healthcare services.

ELIGIBILITY:
Inclusion criteria

* Experts in cardiology
* Experts in personalized medicine
* Experts in digital health.

Exclusion criteria

- Failure to provide informed consent (i.e., non-acceptance of the informed consent form)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A panel of at least 10 experts will be recruited from professionals involved in the INNOPREV project (internal and/or external members) with expertise in cardiology, personalized medicine, and/or digital health. Participation will be by email invitation and will require acceptance of the informed consent form (exclusion criterion: failure to provide informed consent)
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Achievement of expert-panel consensus on recommendations for the implementation of PRS and wearable devices, as assessed by the Content Validity Index (CVI) | At the end of the Delphi process (up to 4 months)
  Achievement of consensus among the expert panel on the proposed recommendations. Consensus will be defined, for each item, as a Content Validity Index (CVI) > 79%, where the CVI represents the proportion of experts assigning a rating of 4 or 5

SECONDARY OUTCOMES:
Identification of recommendations with partial agreement (CVI 70-79%) | After each Delphi round, through completion of the process (up to 4 months)
  Identification of items/recommendations with a Content Validity Index (CVI) between 70% and 79%, indicating the need for item revision and/or additional Delphi rounds
Development of the final set of recommendations, structured by domain (genomic, digital, and clinical/organizational) | At completion of the Delphi process (up to 4 months)
  Production of the final set of recommendations, organized by domain (genomic, digital, and clinical/organizational)
Stability of responses across successive rounds (assessment of changes in CVI) | Between successive Delphi rounds, until completion of the process (up to 4 months)
  Assessment of response stability by comparing, for each item, changes in the CVI across successive Delphi rounds

CONTACTS AND LOCATIONS:
Overall Officials: STEFANIA BOCCIA, PHD, Principal Investigator — Policlinico Universitario Fondazione Agostino Gemelli IRCCS
Locations (1):
- Policlinico Universitario Fondazione Agostino Gemelli IRCCS, Roma, RM, Italy